CLINICAL TRIAL: NCT03400462
Title: Comparison of the Effectiveness of Three Different Treatment Methods in Myofascial Pain Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Principal Investigator, Dalewski Bartosz, DMD, PhD, Pomeranian Medical University Szczecin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KB-0012/83/16
Record Dates: First submitted 2018-01-01; First posted 2018-01-17 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Temporomandibular Disorder
Keywords: Dry needling, occlusal splint, NSAID, nimesulide
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Anti-Inflammatory Agents, Non-Steroidal; Dry Needling

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- dry needling + oral appliance (Experimental): Three visits are needed in this therapy method. Visits schedule:( 1st visit - Day 1st , 2nd visit- 7 days after the 1st, 3rd visit- 7 days after the 2nd) Equipment: acupuncture needle 0,6*13 e.g. Dragon Medical Device, solution for skin disinfection, sterile gauze. Exposition time : 30 minutes once a week
  Interventions: Device: oral appliance; Other: dry needling
- antiinflammatory drugs + splint therapy (Experimental): Patient's instruction for NSAID use:
  Nimesulide 2*100 mg/ 24 h- twice a day one pill of the 100 mg Nimesulide during 14 days
  Interventions: Drug: NSAID; Device: oral appliance
- splint therapy (Active Comparator): Splint therapy is an useful treatment method for several group of patients e.g TMD patients, patients with retrodiscitis, patients with muscle pain disorders like local muscle soreness or chronic myalgia.
  The patients have been instructed to use the appliance during nighttime. After 7 days the patient had to came back for a control visit.
  Interventions: Device: oral appliance

INTERVENTIONS:
Drug: NSAID — Nimesulide has anti-inflammatory and analgesic properties. Like other NSAIDs it inhibits the action of COX . If prostaglandins can not be further synthesized, so there is no factor able to excite local nociceptors. According to t must be taken regularly for a minimum 2 weeks to achieve appropriate blood concentration.
  Other Names: nimesulid
  Arms: antiinflammatory drugs + splint therapy
Device: oral appliance — The stabilization appliance used in this study was a removable device for maxillary arch, made of hard acrylic. Appliance was fitted over occlusal and incisal surfaces of the teeth and precisely contacted with the teeth of opposing arch. It provided canine disocclusion of the posterior teeth during eccentric movements.
Other: dry needling — Equipment: acupuncture needle 0,6*13 e.g. Dragon Medical Device, Visits schedule:( 1st visit - Day 1st , 2nd visit- 7 days after the 1st, 3rd visit- 7 days after the 2nd)
  Arms: dry needling + oral appliance

SUMMARY:
The aim of this study was to compare the effectiveness of myofascial pain treatment methods.

DETAILED DESCRIPTION:
Three different metoda were taken into account: dry needling, occlusal sprint therapy and NSAID therapy.

ELIGIBILITY:
Inclusion Criteria:

* pain localized in the TMJ or in the preauricular area.
* no other analgesic treatment in the area of head and neck during last 12 months

Exclusion Criteria:

* inflammation in the oral cavity that emerge as a myofascial pain
* earlier splint therapy
* pharmacotherapy e.g oral contraception, hormone replacement therapy, -antidepressants
* systemic diseases e.g. rheumatic, metabolic
* lack of stability in the masticatory organ motor system
* masticatory organ injury

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-12-12 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 6 months
  It is a continuous scale comprised of a horizontal line, usually 10 cm in length. "no pain" (score of 0) and "pain as bad as it could be (score of 10)

CONTACTS AND LOCATIONS:
Overall Officials: Bartosz Dalewski, DMD,PhD, Principal Investigator — Pomeranian Medical University

IPD SHARING:
Plan to Share IPD: Undecided